CLINICAL TRIAL: NCT06398275
Title: Remimazolam for Emergence Delirium Prevention in Patients Undergoing Rhinoseptoplasty, FESS or Septoplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Grgur Prižmić, MD, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 520-03/24-01/14
Record Dates: First submitted 2024-04-29; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-01

CONDITIONS: Remimazolam; Emergence Delirium; Rhinoplasty
Keywords: Remimazolam
MeSH Terms: conditions — Emergence Delirium | interventions — remimazolam; Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Remimazolam 20 MG Injection [Byfavo]
- 2 (Placebo Comparator)
  Interventions: Drug: NaCl 0.9%

INTERVENTIONS:
Drug: Remimazolam 20 MG Injection [Byfavo] — Remimazolam 0.1 mg/kg intravenous injection
  Arms: 1
Drug: NaCl 0.9% — NaCl 0.9% 0.04 mL/kg
  Arms: 2

SUMMARY:
The aim of this research is to confirm the effectiveness of remimazolam in preventing delirium during recovery from anesthesia in adult patients who have undergone one of the rhinological surgeries (septoplasty, rhinoseptoplasty or functional endoscopic sinus surgery).

Patients aged 18-65, ASA classification I-II will be anesthetized with balanced anesthesia maintained with sevoflurane and will be randomized into two groups. The first group will receive remimazolam before anesthesia, while the second will receive normal saline solution.

The main outcome of the study will be the presence/absence of delirium during anesthesia recovery, while the secondary outcome will be the postoperative pain level, the length of stay in the recovery room, the presence of unwanted events in the recovery room, and the presence of postoperative mood changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for rhinoplasty, rhinoseptoplasty or FESS
* ASA I or II

Exclusion Criteria:

* pregnancy
* patients treated with psychiatric medication (in the time of operation or 6 months prior to operation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Richmond agitation sedation scale | Immediately after extubation and every five minutes after that for half hour

CONTACTS AND LOCATIONS:
Locations (1):
- UH Split, Split, Croatia